CLINICAL TRIAL: NCT07138755
Title: The Efficacy and Safety of the Combination of Sintilimab With Platinum-doublet Chemotherapy and Adaptive Radiotherapy Strategy in the Treatment of Stage III Non-small Cell Lung Cancer Patients
Brief Title: The Efficacy and Safety of the Combination of PD-1 With Chemotherapy and Adaptive Radiotherapy Strategy in the Treatment of Stage III Non-small Cell Lung Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Xuewen Liu, Professor, The Third Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R25063
Record Dates: First submitted 2025-07-24; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: NSCLC; Sintilimab; Adaptive Radiotherapy
Keywords: V20; stage III NSCLC; Adaptive Radiotherapy; sintilimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adaptive radiotherapy strategy (Experimental): After two cycles of sintilimab and platinum based chemotherapy, receive two additional courses of sintilimab and platinum based chemotherapy and adaptive radiotherapy strategy
  Interventions: Drug: Experimental

INTERVENTIONS:
Drug: Experimental — Drug: Sintilimab, 200mg IV D1 Q3W, Cisplatin, 75mg/m2 D1 IV Q3W or Carboplatin AUC 5 D1 IV Q3W, Paclitaxel or Paclitaxel liposome 135-175mg/m2 D1 IV Q3W(Squamous） Drug: Sintilimab, 200mg IV D1 Q3W, Cisplatin, 75mg/m2 D1 IV Q3W or Carboplatin AUC 5 D1 IV Q3W, Pemetrexed, 500mg/m2 D1 IV Q3W(adenocarcinoma） Radiation:Adaptive radiotherapy with V20<20%: 1.PGTV60-66Gy/2.0-2.2Gy/30F;PTV54Gy/1.8Gy/30F;2.PGTV54-66Gy/2.0-2.2Gy/30F；3.PGTV50Gy/2.0Gy/25F

SUMMARY:
To evaluate the Efficacy and Safety of the Combination of Sintilimab With Platinum-doublet Chemotherapy and Adaptive Radiotherapy Strategy in the Treatment of Stage III Non-small Cell Lung Cancer Patients

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are willing and able to comply with the scheduled visits, treatment plans, laboratory tests, and other requirements of the study
2. Age range of 18-75 years old upon enrollment, both male and female are eligible
3. Stage III NSCLC confirmed by histology or cytology (according to the International Union Against Cancer and the Joint American Committee on Cancer 8th edition TNM staging of lung cancer)
4. It was clarified that surgical resection is not possible After MDT discussion,
5. The main driver genes have no sensitive mutations (including EGFR, ALK, ROS1, MET, HER2, etc.)
6. No previous systematic anti-tumor treatment or chest radiotherapy for NSCLC
7. According to RECIST v1.1, there is at least one measurable lesion, and according to RECIST v1.1, this lesion is suitable for repeated and accurate measurements
8. There is sufficient organ function reserve to meet the needs of clinical research

Exclusion Criteria:

1. There are any small cell carcinoma components present in the histopathology, as well as special types such as salivary gland type and SMARCA4 deficiency
2. Except for NSCLC, the subjects had other malignant tumors within the 5 years prior to enrollment. Subjects with other tumors that have been cured by local treatment, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast cancer in situ, are not excluded
3. Previously received local treatments for tumor lesions such as thoracic radiotherapy and radiofrequency ablation
4. Received non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, tumor necrosis factor, etc., excluding IL-11 used to treat thrombocytopenia) within 2 weeks before the first administration; Received Chinese herbal medicine or traditional Chinese patent medicines and simple preparations with anti-tumor indications within 1 week before the first administration
5. Suffering from active autoimmune diseases that require systematic treatment within the past two years
6. History of immunodeficiency; Individuals who test positive for HIV antibodies; Currently in long-term use of systemic corticosteroids or other immunosuppressants
7. Subjects who are known to have active pulmonary tuberculosis (TB) and suspected of having TB need to undergo clinical examination to exclude them; Known active syphilis infection
8. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
9. Previous or current non infectious pneumonia/interstitial lung disease requiring systemic corticosteroid therapy
10. Serious infection occurred within 4 weeks prior to the first administration, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; Active infections that have received systemic anti infective therapy within 2 weeks prior to the first administration (excluding antiviral therapy for hepatitis B or C)
11. Current active hepatitis B subjects (HBsAg positive and HBV-DNA exceeding 1000 copies/ml (200IU/ml) or above the detection limit)
12. Tumor invasion or compression of important surrounding organs (such as aorta, heart and pericardium, superior vena cava, trachea, esophagus, etc.) or the risk of developing esophagotracheal fistula or esophageal pleural fistula; Tumor mediastinal lymph node metastasis invading the trachea and main bronchus with the risk of bronchial fistula
13. History of myocarditis, cardiomyopathy, and malignant arrhythmia in the past
14. Within 6 months prior to the first administration, there is a history of esophageal and gastric varices, severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding
15. Any arterial thromboembolic event, NCI CTCAE 5.0 grade 3 or higher venous thromboembolic event, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy occurred within 6 months prior to the first administration; Currently, there is hypertension and after treatment with oral antihypertensive drugs, the systolic blood pressure is ≥ 160mmHg or the diastolic blood pressure is ≥ 100mmHg
16. History of severe bleeding tendency or coagulation dysfunction
17. Received a live vaccine within 30 days prior to the first administration, or planned to receive a live vaccine during the study period
18. Known to be allergic to any component of any anti-tumor drug; Known history of severe hypersensitivity reactions to other monoclonal antibodies
19. Known history of mental illness, drug abuse, alcoholism, or drug use
20. Pregnant or lactating women
21. Any past or current diseases, treatments, or laboratory abnormalities that may confuse the research results, affect the participants' full participation in the study, or may not be in the best interests of the participants
22. Local or systemic diseases caused by non malignant tumors, or diseases or symptoms secondary to tumors, which can lead to higher medical risks and/or uncertainty in survival evaluation, such as tumor like leukemia reactions (white blood cell count>20 × 109/L), cachexia manifestations (such as known weight loss of more than 10% in the first 3 months of screening), etc

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 28 months
  The time from the beginning of treatment to the time when the disease progresses or the patient dies from any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 28 months
  the rate of patients with PR and CR
Disease Control Rate (DCR) | 28 months
  the rate of patients with PR and CR and SD
Overall Survival (OS) | 28 months
  The time from the beginning of treatment to the time when the patient dies from any cause
AE | 28 months
  Incidence of Treatment-Emergent Adverse Events

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/39489090/